CLINICAL TRIAL: NCT06905860
Title: Intra-articular Infiltration of Platelet-Rich Fibrin vs Corticosteroid in Mild to Moderate Knee Osteoarthritis
Acronym: iPRF
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rodrigo de Almeida Mastrorosa, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 75935723.4.0000.5505
Record Dates: First submitted 2025-02-04; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Gonarthrosis; Primary
Keywords: gonarthrosis; i-PRF
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Randomized double-blind clinical trial comparing intra-articular injection of PRF versus intra-articular injection of corticosteroids in mild to moderate arthrosis of the knee. Inclusion criteria: Age 50 years or older, who have not improved with non-surgical treatment for at least 3 months, ability to sign informed consent, mean visual analogue scale > 40/100 (over at least 7 days during the month anterior), mild or moderate knee arthrosis diagnosed by grade 2 or 3 radiographic imaging according to the Kellgren-Lawrence classification. Inclusion criteria: angular deviation >10º of varus or valgus in relation to the anatomical neutral axis in the coronal plane clinically evaluated with a goniometer (femur anatomical axis x tibial anatomical axis > 4th varus or > 16th valgus), BMI >35 or <18, smoking , autoimmune inflammatory disease - rheumatologic, diabetes - with glycated Hb > 7, chronic kidney disease, coagulopathies, severe cardiovascular diseases, infections or immunodeficiencies,
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding after the assignment of patients to their groups will be carried out as follows:
  Participants: Blinding. Both the intervention group and the control group will receive the same preparations, undergo the same blood collections, and be subjected to infiltration intervention.
  Investigators: Blinding. Only the person responsible for opening the envelopes will know to which group each patient was allocated. The investigators will only know the group of each patient after the statistical analysis is completed.
  Intervention providers: Blinding. Only the person responsible for opening the envelopes will know to which group each patient was allocated.
  Data recorders: Some data will be collected in person by individuals who will not have access to information about which group each patient belongs to, as only the person responsible for opening the envelopes will know in which group each patient was allocated. Some data will be collected remotely.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Corticoid (Active Comparator): The procedures will be performed by the same doctor. The patients will be blinded so that they do not know to which group each individual belongs. In this group, 40ml of peripheral blood will also be collected and placed for centrifugation. During the preparation for the application, a nurse (who will not participate in the study) will have a list of the randomization and will prepare the material in an opaque syringe (blinding both the applicator and the patient).
  In this group of patients, a solution of 10ml containing 40mg of Triamcinolone will be administered in the first application and 10ml of saline in the second and third applications, with intervals of 14 to 28 days between the applications. The applications will be performed on an outpatient basis, with patients being advised to follow the same protocol for physiotherapy and rehabilitation. There will be no restrictions on load or range of motion in the knee being treated.
  Interventions: Drug: Corticosteroid
- platelet-rich fibrin (Experimental): The Intervention Group consists of the intra-articular application of PRF in the knee. The applications will be performed by the same doctor. The patients will be blinded so that they do not know to which group each individual belongs. A total of 3 applications of PRF will be conducted, with intervals of 14 to 28 days between them.
  10ml of PRF will be applied intra-articularly, on an outpatient basis, with patients being instructed to follow the same protocol for physiotherapy and rehabilitation. There will be no restrictions on load or range of motion in the knee being treated.
  Interventions: Drug: Platelet-rich fibrin (PRF)

INTERVENTIONS:
Drug: Platelet-rich fibrin (PRF) — The Intervention Group consists of the intra-articular application of PRF in the knee. The applications will be performed by the same doctor. The patients will be blinded so that they do not know to which group each individual belongs. A total of 3 applications of PRF will be conducted, with intervals of 14 to 28 days between them.
  10ml of PRF will be applied intra-articularly, on an outpatient basis, with patients being instructed to follow the same protocol for physiotherapy and rehabilitation. There will be no restrictions on load or range of motion in the knee being treated.
  Arms: platelet-rich fibrin
Drug: Corticosteroid — The procedures will be performed by the same doctor. The patients will be blinded so that they do not know to which group each individual belongs. In this group, 40ml of peripheral blood will also be collected and placed for centrifugation. During the preparation for the application, a nurse (who will not participate in the study) will have a list of the randomization and will prepare the material in an opaque syringe (blinding both the applicator and the patient).
  In this group of patients, a solution of 10ml containing 40mg of Triamcinolone will be administered in the first application and 10ml of saline in the second and third applications, with intervals of 14 to 28 days between the applications. The applications will be performed on an outpatient basis, with patients being advised to follow the same protocol for physiotherapy and rehabilitation. There will be no restrictions on load or range of motion in the knee being treated.
  Other Names: corticoid
  Arms: Corticoid

SUMMARY:
Methodology: Randomized double-blind clinical trial comparing intra-articular injection of Platelet-Rich Fibrin (PRF) versus intra-articular injection of corticosteroids in mild to moderate arthrosis of the knee. Inclusion criteria: Age 50 years or older, who have not improved with non-surgical treatment for at least 3 months, ability to sign informed consent, mean visual analogue scale > 40/100 (over at least 7 days during the month anterior), mild or moderate knee arthrosis diagnosed by grade 2 or 3 radiographic imaging according to the Kellgren-Lawrence classification. Inclusion criteria: angular deviation >10º of varus or valgus in relation to the anatomical neutral axis in the coronal plane clinically evaluated with a goniometer (femur anatomical axis x tibial anatomical axis > 4th varus or > 16th valgus), BMI >35 or <18, smoking , autoimmune inflammatory disease - rheumatologic, diabetes - with glycated Hb > 7, chronic kidney disease, coagulopathies, severe cardiovascular diseases, infections or immunodeficiencies, malignant neoplasm in activity or under treatment, use of NSAIDs in the last month, use of corticosteroids in the last 3 months, platelets < 150,000, recent intra-articular corticosteroid infiltration or recent Hyaluronic acid infiltration (within the last 6 months), pregnancy or suspected pregnancy, psychiatric disorders. Exclusion criteria: when one of the investigators considers that the participant may be simulating a worse health state than the real one in order to receive financial assistance with the absence from work, he will be excluded from the work. Primary outcome: WOMAC. Secondary outcomes: Visual Analogue Pain Scale. Evaluation moments: inclusion and after the procedure at 3, 6, 12, 18 and 24 months. Sample calculation: 90 patients, 45 patients in each group, considering 15% loss to follow-up and aiming to reach a power of 0.8 and an alpha value of 0.5.

DETAILED DESCRIPTION:
The objective of this work is to compare the efficacy of intra-articular injection of PRF versus intra-articular application of corticosteroid in the treatment of patients with mild to moderate knee osteoarthritis This study will be a prospective, randomized, double-blind, comparative clinical trial with a 1:1 allocation ratio following the CONSORT (Consolidated Standards of Reporting Trials) guidelines. Patients with knee osteoarthritis will be screened at the Knee Outpatient Clinic of the Department of Orthopedics and Traumatology of EPM-UNIFESP.

The Intervention Group consists of intra-articular application of PRF in the knee, while the Control Group consists of intra-articular application of corticosteroids in the knee. For patients in both groups (PRF or corticosteroid), 40ml of venous blood will be collected for the preparation of PRF, and the infiltration will be performed or not, according to random allocation. For patients in the corticosteroid group, the blood sample will be discarded.

The Intervention Group consists of intra-articular application of PRF in the knee. The applications will be performed by the same physician. Patients will be blinded to ensure they do not know which group each individual belongs to. Three applications of PRF will be carried out with intervals of 14 to 28 days between them.

A total of 10ml of PRF will be applied intra-articularly, on an outpatient basis, with patients being instructed to follow the same physical therapy and rehabilitation protocol. There will be no restrictions on weight-bearing or range of motion in the knee during the application. As a rescue medication for pain, if VAS > 3, patients may use Paracetamol 750mg every 6 hours per day and/or Dipyrone up to 1g every 6 hours per day. If they experience VAS > 7, they may use Tramadol 100mg every 6 hours, with all medications being monitored.

The procedures will be performed by the same doctor. The patients will be blinded so that they do not know to which group each individual belongs. In this group, 40ml of peripheral blood will also be collected and placed for centrifugation. During the preparation for the application, a nurse (who will not participate in the study) will have a list of the randomization and will prepare the material in an opaque syringe (blinding both the applicator and the patient).

In this group of patients, a solution of 10ml containing 40mg of Triamcinolone will be administered in the first application and 3ml of saline in the second and third applications, with intervals of 14 to 28 days between the applications. The applications will be performed on an outpatient basis, with patients being advised to follow the same protocol for physiotherapy and rehabilitation. There will be no restrictions on load or range of motion in the knee being treated. As rescue medication for pain, if the Visual Analog Scale (VAS) score is greater than 3, patients may use Paracetamol 750mg every 6 hours per day and/or Dipyrone up to 1g every 6 hours per day. If they have a VAS score greater than 7, they may use Tramadol 100mg every 6 hours, with all medications being monitored.

The assessments will include the Visual Analog Scale for Pain and the WOMAC questionnaire. The primary outcome will be the WOMAC (Pain subscale). The average time to complete these questionnaires is 10 minutes. All outcomes will be assessed at the time of inclusion in the study and after the procedure at 3 months, 6 months, 12 months, 18 months, and 24 months. All patients will also be evaluated 2 weeks after the procedure to investigate possible complications. Additionally, evaluations of other secondary outcomes such as physiotherapy participation, amount of analgesic use, and knee range of motion will be conducted.

The questionnaires will be sent and answered by patients electronically, and the analyses will be carried out by a statistician. Patients and statisticians performing the assessments and analyses will be blinded to each task so that they do not know to which group each individual belongs.

A clinical failure will be considered if a patient's pain is greater than or equal to the pain they experienced before the interventions, occurring more than 50% of the days in the last month or assessment period (the period between evaluations). These failures will be reported as efficacy over 6 months, 1 year, and 2 years. Based on these results, the patient may undergo another treatment (which could be the same treatment they previously received or not).

ELIGIBILITY:
Inclusion Criteria:The following inclusion criteria will be followed:

* Age 50 years or older
* Who have not improved with non-surgical treatment for at least 3 months, ability to sign a consent form, average visual analog scale > 40/100 (over at least 7 days in the previous month)
* Mild or moderate knee osteoarthritis diagnosed by radiographic imaging grade 2 or 3 according to the Kellgren-Lawrence classification.

Exclusion Criteria: The exclusion criteria will be:

-Absence from work due to disability benefits or income reduction assistance (worker's compensation). Whenever one of the investigators believes that a participant may be simulating a worse health condition than reality to receive financial assistance with work absence, they will be excluded from the study.

The following non-inclusion criteria will be observed:

* Angular deviation >10º of varus or valgus in relation to the anatomical neutral axis in the coronal plane assessed clinically with a goniometer (anatomical axis of the femur x anatomical axis of the tibia > 4º varus or > 16º valgus)
* Body Mass Index (BMI)>35 or <18
* Smoking
* Autoimmune inflammatory disease - rheumatological
* Diabetes - with HbA1c > 7
* Chronic kidney disease
* Coagulopathies
* severe cardiovascular diseases
* infections or immunodeficiencies
* active or treated malignant neoplasia
* use of NSAIDs in the last month
* use of corticosteroids in the last 3 months
* platelets < 150,000
* recent intra-articular corticosteroid injection or recent HA injection (in the last 6 months)
* pregnancy or suspected pregnancy
* psychiatric disorders.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | All outcomes will be evaluated at the time of inclusion in the study and after the procedure at 3 months, 6 months, 12 months, 18 months, and 24 months
  The following will be assessed: Western Ontario and McMaster Universities Arthritis Index (WOMAC) 0-100. The primary outcome will be WOMAC Pain subscale. The average time to complete these questionnaires is 10 minutes. All outcomes will be evaluated at the time of inclusion in the study and after the procedure at 3 months, 6 months, 12 months, 18 months, and 24 months. All patients will also be evaluated 2 weeks after the procedure to investigate possible complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data sharing is essential for scientific transparency, study reproducibility, and the advancement of knowledge. However, it is crucial to protect participants' privacy, especially when the data contains sensitive information. The study data will be submitted for publication in a scientific journal after anonymization
  Regarding the data, its handling, treatment, protection, confidentiality, and transparency, the Data Management Plan Tool - DMPTOOL (https://dmptool.org/) will be used, with institutional identification from UNIFESP. One of the researchers involved will access DMPTOOL through their UNIFESP institutional email to create the data management plan for this project, which will be submitted to the UNIFESP Dataverse research data repository (https://repositoriodedados.unifesp.br).
Supporting Information: SAP, CSR
Time Frame: Data will be released after 2 years of patient follow-up, and will remain available for 5 years
Access Criteria: After the study is completed, the data may be shared with researchers affiliated with universities. Each request will be assessed individually by the principal investigator and the data will be released for access on the linked research website.
URL: https://repositoriodedados.unifesp.br